CLINICAL TRIAL: NCT06249100
Title: Flexible Mini Percutaneous Nephrolithotomy Vs Retrograde Intra-renal Surgery for Treatment of Renal Stones: a Randomized Controlled Trial
Brief Title: Flexible Mini Percutaneous Nephrolithotomy Vs Retrograde Intra-renal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 351/2023
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-07

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- flexible mini percutaneous nephrolithotomy (Experimental): In Group A (flexible mini-PCNL cases), puncture will be done under fluoroscopic guidance medial to the posterior axillary line using an 18-gauge puncture needle. The puncture will be directed horizontally or with slight upward inclination towards lower or middle calyx. After a successful puncture, a 0.035 Fr Super Stiff guidewire will be inserted either to the ureter or to another calyx. Tract dilatation will be done with Storz 15/16 Fr one step metal dilator followed by 16.5 Fr access sheath. Stone disintegration will be done with the flexible mini-nephroscopy (WiScope Digital Endoscope System by OTU Medical, California, USA) which has a shaft length of 38 cm, distal tip diameter is 15.3 F tapering to 10 F, working channel inner diameter is 6.6 F, and the angle of deflection of distal tip is 210 degrees.
  Interventions: Procedure: flexible mini percutaneous nephrolithotomy
- retrograde intrarenal surgery (Active Comparator): In Group B (retrograde intrarenal surgery cases), a 0.035 Fr guidewire will be inserted into the ureteric orifice under fluoroscopic guidance. Ureteric dilatation will be done with serial semi-rigid dilators 6- 16 Fr (Nidhi Meditech) followed by 14-16 Fr access sheath. Stone disintegration will be done with the LithoVue Flexible URS (Boston Scientific, Massachusetts, U.S.) which has a shaft length of 68 cm, distal tip diameter is 7.7-10 F, working channel inner diameter is 3.6 F, and the angle of deflection of distal tip is 270 degrees.
  Interventions: Procedure: Retrograde intrarenal surgery

INTERVENTIONS:
Procedure: flexible mini percutaneous nephrolithotomy — In Group A (flexible mini-PCNL cases), a puncture will be done under fluoroscopic guidance medial to the posterior axillary line using an 18-gauge puncture needle. The puncture will be directed horizontally or with a slight upward inclination towards the lower or middle calyx. After a successful puncture, a 0.035 Fr Super Stiff guidewire will be inserted. Tract dilatation with amplatz dilator followed by access sheath insertion. Stone disintegration will be done with the flexible mini-nephroscopy (WiScope Digital Endoscope System by OTU Medical, California, USA) which has a shaft length of 38 cm, distal tip diameter is 15.3 F tapering to 10 F, working channel inner diameter is 6.6 F, and the angle of deflection of the distal tip is 210 degrees.
  Arms: flexible mini percutaneous nephrolithotomy
Procedure: Retrograde intrarenal surgery — n Group B, Flexible ureteroscopy will be used with a ureteral access sheath and laser fragmentation of renal stones will be done
  Arms: retrograde intrarenal surgery

SUMMARY:
The use of flexible ureteroscopy and minimally-invasive percutaneous techniques, which utilize smaller tract sizes, has been established as a way to decrease the invasiveness of procedures and improve patient outcomes compared to conventional percutaneous nephrolithotomy (PCNL) and flexible mini-PCNL has emerged as a novel technique previously first as an auxiliary procedure and then as a standalone technique. This study aims to assess the feasibility and effectiveness of flexible nephoscopy in improving stone clearance compared to standard retrograde intrarenal surgery using a flexible ureteroscope.

DETAILED DESCRIPTION:
Urinary stones are one of the most common rising health concerns around the world. Urolithiasis is particularly common in high-income countries, with more than 10% of people suffering from it. Renal stones often manifest as colicky loin pain, often known as renal colic.

Percutaneous nephrolithotomy (PCNL) is highly recommended by international guidelines as the primary treatment for renal stones larger than 20 mm. However, for stones ranging from 10 to 20 mm in size, treatment options may include shock wave lithotripsy (SWL), PCNL, or retrograde intrarenal surgery (RIRS).

Significant advancements have been achieved in surgical techniques recently, leading to the emergence of minimally invasive percutaneous nephrolithotomy (mini-PCNL) as a viable and effective treatment option for the removal of large renal and proximal ureteral stones.

In recent years, there has been a consistent reduction in the size of endoscopic instruments. The primary objective of these tools is to minimize the amount of blood lost during surgery, lower the occurrence of complications both during and after the operation, and ultimately reduce the length of hospital stays.

Despite the use of a smaller nephroscope, the rigidity of the mini-nephroscope poses a limitation in maneuvering into renal calyces at acute angles. This limitation may necessitate the creation of additional tracts, leading to an increase in morbidity. To tackle this challenge, a new technique flexible mini-nephroscope has been developed. This innovative instrument allows for access to all regions of the pelvi-caliceal system through a single access tract.

Retrograde Intrarenal Surgery (RIRS) is a prominent approach utilized to eliminate kidney stone disease. In contrast to PCNL, RIRS offers the benefit of utilizing a natural orifice, thereby eliminating the need for an additional pathway for lithotripsy. Consequently, this treatment option ensures enhanced safety and facilitates a more favorable postoperative recovery process.

RIRS has some significant limitations that make it challenging to retrieve a large number of fragments after the lithotripsy of large stones. Additionally, there is a complicated balance between irrigation and intrarenal pressure that must be maintained. While continuous rinsing of renal cavities is necessary to improve visibility, an imbalanced fluid evacuation can lead to a rise in pressure within the collecting system. Due to these limitations, large stones cannot be treated with a single RIRS procedure, and multiple sessions may be required. This exposes the patient to repeated anesthesia and the risk of ureteral damage and stenosis, making it important to limit operative time and prevent complications.

This study aims to compare the clinical outcome in the form of safety and efficacy between flexible mini-nephroscopy in minimally-invasive PCNL and retrograde intra-renal surgery in patients with symptomatic renal stones.

ELIGIBILITY:
Inclusion Criteria:

* All patients above the age of 16 years of either sex presented to the Urology clinic in our university hospitals
* kidney stones with a size not exceeding 3.0 cm (estimated by CTUT as the greatest dimension or the summation of the greatest dimensions in case of more than one stone detected)

Exclusion Criteria:

* Patients with lumber hernia on the same site of the surgery
* Patients with a stone burden exceeding 3cm
* Patients with renal anomalies preventing access
* Patients with coagulopathies/bleeding tendency
* Patients with untreated or active UTI

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
stone-free rate | 1 month postoperative
  patients will be considered stone free, if the stone residual in the follow up is less than 4mm

SECONDARY OUTCOMES:
Operative time | 24 hour postoperative
  time from starting the procedure with the cystoscopy till termination with catheter insertion. intraoperative finding in minutes
Hospital Stay | 1 month postoperative
  duration of hospital stay since admission on the day of the procedure till discharge
Cost analysis | 1 month postoperative
  evaluation of the procedure cost, the additional cost of hospital stay, complication and auxiliary procedure needed for stone residual.
infection rate | up to 1 month postoperative
  evaluation of postoperative urinary tract infection
Hemoglobin drop | 1 day postoperative
  evaluation of hemoglobin drop in the procedure by CBC

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No